CLINICAL TRIAL: NCT05897931
Title: Effects of Connective Tissue Massage and Taping in Patients With Fibromyalgia
Brief Title: Effects of Two Different Applications in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Eylül Pınar KISA, assistant professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fibromyalgia
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective tissue massage (Experimental): Participants will receive TENS and infrared treatment for 25 minutes, 5 days a week. Then Connective Tissue Massage will be applied.
  Interventions: Other: Connective tissue massage
- Kinesio Tape Application (Experimental): Participants will receive TENS and infrared treatment for 25 minutes, 5 days a week. Kinesio tape application will be applied 2 days a week for 4 weeks.
  Interventions: Other: Kinesio Tape Application

INTERVENTIONS:
Other: Connective tissue massage — Connective Tissue Massage will be applied by starting from the lumbosacral region, continuing from the lower thoracic region, and finishing by applying it to the scapular region, interscapular region, and cervico-occipital region.
  Arms: Connective tissue massage
Other: Kinesio Tape Application — Taping will be applied to the levator scapula and upper trapezius muscles in a "Y" shape, with 25% tension and while the participants were in an upright position. Again in the same position, this time the "C" shaped taping technique will be adhered with 50% tension from the middle fibers of the trapezium to the last rib.
  Arms: Kinesio Tape Application

SUMMARY:
The study aims to determine the effect of connective tissue massage and taping applications on the pain and depression complaints of fibromyalgia patients and to compare their impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with fibromyalgia.
* Be in the age range of 20 - 55 years.
* To be a volunteer participant in the research.
* Being able to communicate comfortably.
* To be able to act independently.

Exclusion Criteria:

* Having had a surgical operation within the last year.
* Presence of significant infection.
* Being diagnosed with cancer.
* Being pregnant or breastfeeding.
* Being addicted to drugs or alcohol.
* Having a cognitive problem.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 4 weeks
  Visual Analogue Scale (VAS) will be used to assess pain severity. In the assessment, the patient is asked to mark pain intensity on a 10-centimeter line that no pain is 0, and the most severe pain is 10.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire | 4 weeks
  The questionnaire assesses the functional status of patients with fibromyalgia. The scale consists of 20 questions that measure physical function, well-being, difficulty in doing work, not being able to go to work, fatigue, stiffness, morning fatigue, pain, anxiety, and depression separately. Low scores indicate improvement or less effect in patients.
McGill Pain Questionnaire | 4 weeks
  The quality of the pain felt by the patients will be evaluated with the Short Form McGill Pain Questionnaire. The level of severity felt by the patient is evaluated with a number scale (0=no, 1=mild, 2=moderate, 3=severe), and higher scores show severe pain intensity.
Beck's Depression Inventory | 4 weeks
  The Beck's Depression Inventory (BDI) is a 21-item self-assessment scale that evaluates the patients' perceived depressive symptoms quantitatively and measures the symptoms of depression. The higher scores indicate the severity of the patient's depression. It has been suggested that those who score 17 and above on the BDI may constitute an at-risk group.
Short Form-36 Quality of Life Scale | 4 weeks
  The scale assesses the quality of life. The scale consists of 36 items evaluated in 8 separate subscales. The score from each subscale is between 0-100, and a higher score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Rasmi Muammer, PhD, Study Chair — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No